CLINICAL TRIAL: NCT01357655
Title: An Open-Label, Randomized, Multicenter Phase 2 Trial of Dasatinib (SPRYCEL®) vs. Dasatinib Plus Smoothened Antagonist (BMS-833923) in the Treatment of Subjects With Newly Diagnosed Chronic Phase Philadelphia Chromosome Positive Chronic Myeloid Leukemia (CML).
Brief Title: Phase 2 Dasatinib Combo With Smoothened (SMO) Antagonist (BMS-833923)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled in this trial could receive the SMO antagonist as a recommended phase 2 dose was not determined by a different, concurrently-run trial.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA180-363; 2011-000083-10 (EudraCT Number)
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-01

CONDITIONS: Leukemia
Keywords: Myelogenous; Chronic; BCR-ABL Positive
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome | interventions — Dasatinib; BMS-833923

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Dasatinib (Active Comparator)
  Interventions: Drug: Dasatinib
- Arm2: Dasatinib + BMS-833923 (Experimental): Dasatinib for 1 year followed by dasatinib plus BMS-833923 for 2 years followed by dasatinib alone for approximately 2 years; depending on response
  Interventions: Drug: Dasatinib; Drug: BMS-833923

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 100 mg, Once daily, approximately 5 years depending on response
  Other Names: Sprycel®
Drug: BMS-833923 — Capsules, Oral, dose to be determined, Once daily, approximately 2 years depending on response
  Arms: Arm2: Dasatinib + BMS-833923

SUMMARY:
The purpose of the study is to compare response rates in newly diagnosed Chronic Phase (CP) CML subjects treated with dasatinib plus BMS-833923 versus dasatinib alone.

DETAILED DESCRIPTION:
1. Design:

   Study Design and Duration as current described are no longer applicable since enrollment was prematurely concluded due to a decision by the sponsor. Subjects currently enrolled in the trial will continue to receive dasatinib alone at a starting dose of 100 mg QD for:
   1. a maximum of 5 years after entry into the study
   2. until progression by Investigators determination/judgment
   3. intolerance to Dasatinib
   4. the study is terminated due to safety concerns or
   5. other administrative reasons as communicated by the sponsor
2. Research Hypothesis :

The research hypothesis and primary objective of this study as originally designed are no longer applicable as subjects enrolment has been terminated due to administrative reasons by the sponsor. The objective of the altered design of this study is to describe the safety profile and tolerability of dasatinib

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age who have signed informed consent
* Philadelphia positive Chronic Myeloid Leukemia (CML) in chronic phase
* Previously untreated chronic phase CML, except for Anagrelide or Hydroxyurea.
* Eastern Co-Operative Group (ECOG) Performance Status (PS) Score 0 - 2

Exclusion Criteria:

* Known Abl-kinase T315I or T315A mutation
* Serious or uncontrolled medical disorder (including infection or cardiovascular disease) or dementia or other serious psychiatric condition
* Prior chemotherapy.
* Women who are pregnant or breastfeeding or Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy during the entire study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (23):
- United States (3):
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Tennessee Oncology Pllc, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Local Institution, San Miguel de Tucumán, Tucumán Province, Argentina
- Belgium (2):
  - Local Institution, Antwerp
  - Local Institution, Bruges
- Local Institution, Edmonton, Alberta, Canada
- Local Institution, Helsinki, Finland
- France (7):
  - Local Institution, Nantes, Cedex
  - Local Institution, Bordeaux
  - Local Institution, Le Chesnay
  - Local Institution, Lille
  - Local Institution, Paris
  - Local Institution, Strasbourg
  - Local Institution, Toulouse
- Poland (5):
  - Local Institution, Chorzów
  - Local Institution, Gdansk
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Wroc#aw
- Spain (3):
  - Local Institution, Madrid
  - Local Institution, Oviedo
  - Local Institution, Pamplona

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 70 participants were enrolled, 66 were treated. Reasons for non-treatment include 1 adverse event and 3 no longer met study criteria. Participants enrolled were only treated with Dasatinib. The Dasatinib + SMO antagonist (BMS-833923) arm did not have participants because the recommended phase 2 dose of the SMO antagonist had not been determined.
Groups:
- Dasatinib: Dasatinib: Tablets, Oral, 100 mg, were given once daily for approximately 1 year before the study was terminated.
- Dasatinib + SMO Antagonist (BMS-833923): No participants were randomized to this arm because no recommended phase 2 dose of the SMO antagonist could be determined (in a separate trial).
  Dasatinib for 1 year followed by dasatinib plus SMO antagonist (BMS-833923) for 2 years followed by dasatinib alone for approximately 2 years; depending on response Dasatinib: Tablets, Oral, 100 mg, Once daily BMS-833923: Capsules, Oral, dose to be determined, Once daily, approximately 2 years depending on response
Period: Overall Study
Arm/Group | Dasatinib | Dasatinib + SMO Antagonist (BMS-833923)
Started | 66 | 0
Completed | 0 | 0
Not Completed | 66 | 0
Not completed — Administrative Reason by Sponsor | 45 | 0
Not completed — Adverse Event Unrelated to Study Drug | 3 | 0
Not completed — Disease Progression | 1 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Maximum Clinical Benefit | 2 | 0
Not completed — Reason Unspecified | 1 | 0
Not completed — Study Drug Toxicity | 11 | 0
Not completed — Subject Withdrew Consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Treated Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib | Dasatinib + SMO Antagonist (BMS-833923) | Total
Number analyzed (Participants) | 66 | 0 | 66
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 64 years | 54 | 0 | 54
  >=65 years | 12 | 0 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 0 | 27
  Male | 39 | 0 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Molecular Response
Description: Major molecular response (MMR) was assessed using BCR-ABL transcript levels measured by real-time quantitative polymerase chain reaction (qPCR). MMR was defined as a ratio BCR-ABL/ABL ≤0.1% on the international scale (ie, at least 3 log reduction from a standardized baseline value). Number of participants with MMR by timepoint are cumulative.
Time Frame: Baseline up to 12 months
Population: Efficacy Sample: all treated participants with at least one assessment on treatment. Participants enrolled in this trial could not be randomized to the Dasatinib + SMO antagonist arm because no recommended phase 2 dose of the SMO antagonist could be determined (in a separate trial).
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib | Dasatinib + SMO Antagonist (BMS-833923)
Number analyzed (Participants) | 64 | 0
Participants
  Baseline | 1 | 0
  3 Months | 9 | 0
  6 Months | 30 | 0
  12 Months | 34 | 0

2. Secondary Outcome: Complete Molecular Response at Any Time
Time Frame: Baseline to End of study (approximately 48 months)
Population: The study was terminated prior to data collection for this endpoint.
Arm/Group | Dasatinib | Dasatinib + SMO Antagonist (BMS-833923)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression-free Survival, Measured by the Time From Start of Treatment to Progression or Death
Time Frame: Baseline to End of study (approximately 48 months)
Population: The study was terminated prior to data collection for this endpoint.
Arm/Group | Dasatinib | Dasatinib + SMO Antagonist (BMS-833923)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Event-free Survival, Measured by the Time From Start of Treatment to Progression, Death or Treatment Discontinuation
Time Frame: Baseline to End of study (approximately 48 months)
Population: The study was terminated prior to data collection for this endpoint.
Arm/Group | Dasatinib | Dasatinib + SMO Antagonist (BMS-833923)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Transformation-free Survival Measured by the Time From Start of Treatment to Criteria for Accelerated or Blast Phase CML Are Met and Death
Time Frame: Baseline to End of study (approximately 48 months)
Population: The study was terminated prior to data collection for this endpoint.
Arm/Group | Dasatinib | Dasatinib + SMO Antagonist (BMS-833923)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAE), Drug-Related Adverse Event (AE), AE Leading to Discontinuation, and Death
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=having certain, probable, possible, or missing relationship to study drug.
Time Frame: From date of first dose of study treatment up to the date of the last dose plus 30 days (approximately 49 months)
Population: All Treated Participants; Participants enrolled in this trial could not be randomized to the Dasatinib + SMO antagonist arm because no recommended phase 2 dose of the SMO antagonist could be determined (in a separate trial).
Measure: Number; unit: participants
Arm/Group | Dasatinib | Dasatinib + SMO Antagonist (BMS-833923)
Number analyzed (Participants) | 66 | 0
participants
  SAE | 18 |
  Drug-Related AE | 56 |
  Death | 2 |
  AE Leading to Discontinuation | 14 |

ADVERSE EVENTS:
Time Frame: From date of first dose of study treatment up to the date of the last dose plus 30 days (approximately 49 months)
Description: All Treated Participants
  Study Initiated: September 14, 2011 Study Completion: January 26, 2016
Groups:
- Dasatinib: Dasatinib: Tablets, Oral, 100 mg, Once daily, approximately 1 year
Arm/Group | Dasatinib
All-Cause Mortality (participants affected / at risk) | 2/66
Serious Adverse Events (participants affected / at risk) | 18/66
Other Adverse Events (participants affected / at risk) | 60/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=66)
Cardiac failure chronic (Cardiac disorders) | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vaginal abscess (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 2
Myocardial ischaemia (Cardiac disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac failure (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 4
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Urosepsis (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Liver abscess (Infections and infestations) | 1
Volvulus (Gastrointestinal disorders) | 1
Amaurosis fugax (Eye disorders) | 1
Apical granuloma (Gastrointestinal disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hypersensitivity (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=66)
Chest pain (General disorders) | 6
Fatigue (General disorders) | 8
Nasopharyngitis (Infections and infestations) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Anxiety (Psychiatric disorders) | 4
Hypertension (Vascular disorders) | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Pharyngitis (Infections and infestations) | 4
Vomiting (Gastrointestinal disorders) | 13
Constipation (Gastrointestinal disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9
Anaemia (Blood and lymphatic system disorders) | 20
Aspartate aminotransferase increased (Investigations) | 4
Diarrhoea (Gastrointestinal disorders) | 18
Headache (Nervous system disorders) | 27
Pyrexia (General disorders) | 10
Weight increased (Investigations) | 4
Abdominal pain (Gastrointestinal disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 11
Sinusitis (Infections and infestations) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Abdominal pain upper (Gastrointestinal disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 5
Gastroenteritis (Infections and infestations) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Insomnia (Psychiatric disorders) | 6
Nausea (Gastrointestinal disorders) | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 14
Peripheral swelling (General disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 8
Acne (Skin and subcutaneous tissue disorders) | 4
Asthenia (General disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 5

LIMITATIONS AND CAVEATS:
No recommended phase 2 dose of the SMO antagonist was determined (in a separate trial). It was decided to discontinue enrollment and end this trial early. The decision was not made due to any new safety signals for dasatinib or the SMO antagonist.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.